CLINICAL TRIAL: NCT01838005
Title: Conditional Cash Transfers to Increase Uptake of and Retention of PMTCT Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Kinshasa School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 12-1676; 1R01HD075171-01 (NIH)
Record Dates: First submitted 2013-03-22; First posted 2013-04-23 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-01

CONDITIONS: HIV
Keywords: Contingency management; conditional cash transfer; PMTCT; Retention; HIV

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (No Intervention): Routine implementation of the national PMTCT guidelines which are an adaptation of the WHO's "Option A"
- Conditional Cash Transfer (Experimental): Financial incentive to attend regular clinic visits and receive PMTCT care
  Interventions: Behavioral: Conditional cash transfer

INTERVENTIONS:
Behavioral: Conditional cash transfer — Eligible women randomized to the intervention group will receive the standard of care plus small and increasing cash payments, on the condition that they attend scheduled clinic visits on time (+/-5days), accept HIV services, deliver in a health facility, and at six weeks postpartum adhere to prescribed infant prophylactic drugs (cotrimoxazole, extended NVP) and provide blood sample for DNA PCR infant early HIV diagnosis.
  Other Names: Contingency management
  Arms: Conditional Cash Transfer

SUMMARY:
The goals of the proposed study are to: 1) test whether small, increasing cash payments to HIV-infected pregnant women, on the condition that they attend scheduled clinic visits and receive proposed services, will increase the proportion of women who receive the most effective antiretroviral regimen they are eligible for by the time of delivery, and 2) elucidate factors that facilitate or inhibit the uptake and adherence to the PMTCT cascade, and to what extent the conditional cash payment program addresses these factors.

This intervention will be implemented and evaluated within our well-established PMTCT program in Kinshasa, Democratic Republic of Congo (DRC),

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed as HIV-positive
* Pregnant between 28 and 32 weeks of gestation (>27 and <32 completed weeks of pregnancy)
* Intend to stay in Kinshasa through delivery and six weeks postpartum
* Able and willing to participate (provide informed consent)

Exclusion Criteria:

* Women will be excluded from the study if they are severely ill and require extended hospitalization or need to be cared for at a referral hospital out of the PMTCT network

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 433 (Actual)
Dates: Start 2013-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
proportion of women who were adherent to all conditionalities and received the most effective ARV intervention they were eligible to receive and delivered at an affiliated maternity | 6 weeks postpartum
  At each monthly visit starting at randomization (28 weeks), participants will be evaluated for the following conditionalities:
  1. attended the scheduled visit on time (+/- 5 days)
  2. accept HIV status and services proposed to them
  3. return to deliver in the clinic At the end of the follow-up (6 weeks post-partum)the proportion of participants who adhered to all these conditions will be calculated for each study group

SECONDARY OUTCOMES:
Mother to child transmission rate at six weeks and HIV-free survival. | 6 weeks post partum
  Proportion of HIV-exposed infant who tested positive at 6 week postpartum
HIV-free survival at 18 month. | 18 months porstpartum
  Proportion of children born to HIV+ enrolled mothers who are alive and non infected with HIV
Proportion of HIV-exposed infants who at their six week visit received extended Nevirapine (NVP) had a DNA PCR test | 6 weeks Postpartum
  Proportion of infants born to HIV-infected participants who at 6 weeks postpartum are receiving the extended nevirapine prophylaxis and have been tested for HIV

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Yotebieng, MD, Principal Investigator — Ohio State University; Emile W Okitolonda, MD, Principal Investigator — Kinshasa School of Public Health
Locations (1):
- Kinshasa School of Public Health, Kinshasa, Kinshasa, Republic of the Congo

REFERENCES:
- [Result] Yotebieng M, Moracco KE, Thirumurthy H, Edmonds A, Tabala M, Kawende B, Wenzi LK, Okitolonda EW, Behets F. Conditional Cash Transfers Improve Retention in PMTCT Services by Mitigating the Negative Effect of Not Having Money to Come to the Clinic. J Acquir Immune Defic Syndr. 2017 Feb 1;74(2):150-157. doi: 10.1097/QAI.0000000000001219. PMID 27787342
- [Result] Yotebieng M, Thirumurthy H, Moracco KE, Kawende B, Chalachala JL, Wenzi LK, Ravelomanana NL, Edmonds A, Thompson D, Okitolonda EW, Behets F. Conditional cash transfers and uptake of and retention in prevention of mother-to-child HIV transmission care: a randomised controlled trial. Lancet HIV. 2016 Feb;3(2):e85-93. doi: 10.1016/S2352-3018(15)00247-7. PMID 26847230
- [Result] Yotebieng KA, Fokong K, Yotebieng M. Depression, retention in care, and uptake of PMTCT service in Kinshasa, the Democratic Republic of Congo: a prospective cohort. AIDS Care. 2017 Mar;29(3):285-289. doi: 10.1080/09540121.2016.1255708. Epub 2016 Nov 6. PMID 27819151
- [Derived] Saleska JL, Turner AN, Gallo MF, Shoben A, Kawende B, Ravelomanana NLR, Thirumurthy H, Yotebieng M. Role of temporal discounting in a conditional cash transfer (CCT) intervention to improve engagement in the prevention of mother-to-child transmission (PMTCT) cascade. BMC Public Health. 2021 Mar 10;21(1):477. doi: 10.1186/s12889-021-10499-0. PMID 33691667